CLINICAL TRIAL: NCT06880705
Title: A Gender-Affirming Stigma Intervention to Improve Substance Misuse and HIV Risk Among Transgender Women
Brief Title: The Trans-Led Care Study
Acronym: TLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Illinois Institute of Technology (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Arryn Guy, Assistant Professor of Psychology, Illinois Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R00DA055508 (NIH); R00DA055508 (NIH)
Record Dates: First submitted 2025-02-26; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Substance Abuse; Substance Addiction; Substance Use Disorder (SUD); Substance Use (Drugs, Alcohol); Human Immunodeficiency Virus (HIV)
Keywords: Substance misuse; HIV risk; Stigma; Psychological distress; Gender affirmation
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome; Social Stigma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (TAU) (No Intervention): Participants randomized to the control condition will receive treatment-as-usual (TAU), following SAMHSA guidelines for risky alcohol and other drug use and CDC established standards of care for STD/HIV prevention counseling. Participants meeting criteria for risky alcohol, drug use, or sexual behavior will be provided 15-25 minutes of brief counseling including: 1) a discussion that the participants drinking or drug use is more than the recommended limits for safe consumption, and that staying below these limits is important for their health; 2) a discussion of HIV risk-reduction interventions (i.e., consistent condom use, PrEP, ART treatment as prevention); and 3) referral to treatment (i.e., regular screening for HIV/STDs, HIV care, and/or substance use treatment).
- The TLC Program (Experimental): Participants randomized to the TLC Program will receive TAU plus the telehealth, peer-delivered group intervention, "the TLC Program."
  Interventions: Behavioral: The TLC Program

INTERVENTIONS:
Behavioral: The TLC Program — Participants randomized to the TLC Program will receive TAU plus the telehealth, peer-delivered group intervention. The TLC Program was adapted from Acceptance and Commitment Therapy (ACT) - an acceptance and mindfulness-based third wave cognitive behavioral therapy. The intervention will be delivered in a group format with peer facilitators via telehealth using videoconferencing. The protocol covers all six ACT core concepts (i.e., contact with the present, acceptance, defusion, self-as-context, values, and committed action) with tailored examples and exercises focused on gender affirmation, internalized stigma, and substance use. Additional sessions are included defining stigma, how stigma affects physical and sexual health and engagement with healthcare, and values-driven self-care goals of substance use reduction and healthcare engagement. Sessions are approximately 1.5 hours each and are delivered over 12 weeks.
  Arms: The TLC Program

SUMMARY:
This study is testing a new mutual-help group called "the TLC program" for transgender adults who use substances or are recently in recovery. The TLC Program is based on Acceptance and Commitment Therapy or "ACT" which is a type of mental health counseling that focuses on using mindfulness skills to connect a person to their values and improve their mental health. The TLC Program was developed by transgender and gender diverse community members, mental health providers, and researchers.

DETAILED DESCRIPTION:
Transgender (trans) populations are disproportionately impacted by HIV compared to the general population (nearly 1 in 7 trans women are living with HIV; 3.2% of trans men are living with HIV compared to 0.3% in the general U.S. population). Trans people also experience stigma rooted in systems of oppression. To prevent the forward transmission of HIV, public health officials emphasize the need for consistent condom use, regular HIV testing, and linkage to HIV prevention and care services. Stigma, however, interferes with trans individuals' ability to engage in HIV prevention and care due to its negative affects across multiple socioecological levels, including structural policies that constrain resources for trans people, negative community attitudes and prejudicial norms towards trans people, interpersonal discrimination towards trans people resulting in social isolation, and trans individual's psychological and behavioral responses to such stigma and stress. This makes stigma a social and structural determinant of health.

Stigma also plays a significant role in increasing risk for substance misuse among trans adults broadly. Rates of current illicit drug use, cannabis consumption, and/or nonmedical prescription drug use among trans adults are high relative to the U.S. general population (29% vs. 10%, respectively). Heavy alcohol use is also high, with 23% of trans adults consuming alcohol on 11 or more days in the past month Prior research with trans women suggests that unmet gender affirmation needs (i.e., the multitude of ways people receive recognition and support for their gender identity) may lead trans women to seek affirmation in traumatizing and unsafe contexts, such as sex work and sex under the influence of substances. Trans women are also at an increased risk of being targeted for violence, including sexual and physical assault, and substance use is associated with increased risks of victimization.

The Model of Gender Affirmation illustrates that lack of gender affirmation (i.e., the multitude of ways people receive recognition and support for their gender identity) contributes to psychological distress, substance misuse, and HIV risk among trans women. Evidence demonstrates that those who experience stigma report attempts to cope by avoiding or controlling distressing thoughts or feelings (e.g., substance use), which in turn produces greater psychological distress, and interferes with self-care behaviors. Specialized evidence-based interventions delivered in community-based organizations have the potential to reduce the negative effects of internalized stigma on behavioral health.

Acceptance and Commitment Therapy (ACT) is one of the few evidence-based approaches that targets stigma related to a variety of conditions, including substance use disorders and HIV. ACT is a transdiagnostic psychotherapeutic intervention that increases psychological flexibility through mindfulness, acceptance, and behavior change processes. ACT for stigma focuses on the fears, shame, and identification with a stigmatized group that pose a barrier to living a life consistent with one's values. ACT is a promising, but not yet evaluated, intervention to improve stigma among trans adults.

Guided by a community-engaged research approach, we are testing an ACT-based, peer-led, gender affirming mutual-help group (called "the TLC Program") to reduce substance misuse and HIV risk among trans adults. The TLC Program was developed through a needs assessment of adaptations to ACT for integration into community-based organizations serving trans populations. Focus groups and interviews with transgender adults and stakeholders (e.g., organization staff, providers who serve trans clients) identified necessary adaptations. A proof-of-concept test of the TLC Program in an open pilot with (N = 16) trans adults who experienced at least one substance use problem in the past year informed final refinements to the intervention. The TLC Program is now being tested in a randomized controlled feasibility/acceptability trial compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

Eligible transgender adults must:

1. be 18 years of age or older;
2. speak primarily English;
3. live in the U.S.;
4. have a gender identity different from their assumed gender, or sex assigned, at birth;
5. identify as a person of transgender experience;
6. endorse having experienced two or more problem(s) related to alcohol or other drug use within the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Gender Minority Stress and Resilience Scale Internalized Transphobia | Reported at baseline assessment, post-assessment (12 weeks), and follow-up assessment (24 weeks)
  Minimum value = 0, Maximum value = 1, Higher score = worse outcome
Health Care Empowerment Inventory | Reported at baseline assessment, post-assessment (12 weeks), and follow-up assessment (24 weeks)
  Minimum value = 1, Maximum value = 5, Higher score = better outcome
Patient-Reported Outcomes Measurement Information System (PROMIS) | Reported weekly, as well as at baseline assessment, post assessment (12 weeks), and follow-up assessment (24 weeks)
  Measuring psychological distress (depression and anxiety), Minimum value = 1 (per subscale), Maximum value = 5 (per subscale), Higher score = worse outcome
Psychological Flexibility, Multidimensional Psychological Flexibility Inventory (MPFI) | Reported at baseline assessment
  Minimum value = 1 (per subscale), Maximum value = 6 (per subscale), Higher score = worse outcome
The Acceptability of Intervention Measure (AIM) | Reported at post-assessment (12 weeks)
  Minimum value = 1, Maximum value = 5, Higher score = better outcome
Intervention Appropriateness Measure | Reported at post-assessment (12 weeks)
  Minimum value = 1, Maximum value = 5, Higher score = better outcome
Feasibility of Intervention Measure (FIM) | Reported at post-assessment (12 weeks)
  Minimum value = 1, Maximum value = 5, Higher score = better outcome

SECONDARY OUTCOMES:
Substance Use Timeline Followback Interview | Over the past 30 days
HIV Risk Questionnaire | Reported at baseline assessment, post-assessment (12 weeks), and follow-up assessment (24 weeks)
  Participants will be reporting number of sexual partners, types of sexual activities, and various HIV risk factors including condom use, PrEP use, and treatment as prevention

OTHER OUTCOMES:
PTSD Life Events Checklist for DSM-5 | Reported at baseline assessment
  Participants will indicate whether certain difficult or stressful life events they have experienced
Intersectional Discrimination Index (InDI) | Reported at baseline assessment
  Minimum value = 0, Maximum value = 13, Higher score = worse outcome
Access to Gender Affirmation in Healthcare Questionnaire | Reported at baseline assessment, post-assessment (12 weeks), and follow-up assessment (24 weeks)
  Minimum value = 1, Maximum value = 5 Higher score = Better outcome
Need for Gender Affirmation Questionnaire | Reported at baseline assessment, post-assessment (12 weeks), and follow-up assessment (24 weeks)
  Minimum value = 1, Maximum value = 5
Satisfaction with Gender Affirmation Questionnaire | Reported at baseline assessment, post-assessment (12 weeks), and follow-up assessment (24 weeks)
  Minimum value = 1, Maximum value = 5, Higher score = better outcome
City Stress Index | Reported at baseline assessment
  Minimum value = 0, Maximum value = 3, Higher score = worse outcome
PCL-5 | Reported at baseline, post-assessment (12 weeks), and follow-up assessment (24 weeks)
  Minimum value = 0, Maximum value = 4, Higher score = worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois Institute of Technology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided